CLINICAL TRIAL: NCT02050178
Title: A Phase 1b Dose Escalation Study of OMP-54F28 in Combination With Nab-Paclitaxel and Gemcitabine in Patients With Previously Untreated Stage IV Pancreatic Cancer
Brief Title: Dose Escalation Study of OMP-54F28 in Combination With Nab-Paclitaxel and Gemcitabine in Patients With Previously Untreated Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54F28-002
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer; Stage IV Pancreatic Cancer
Keywords: Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — OMP-54F28; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: OMP-54F28, Nab-Paclitaxel and Gemcitabine (Experimental)
  Interventions: Drug: OMP-54F28, Nab-Paclitaxel and Gemcitabine

INTERVENTIONS:
Drug: OMP-54F28, Nab-Paclitaxel and Gemcitabine

SUMMARY:
This is an open-label Phase 1b dose-escalation study to assess the safety, tolerability, and PK of OMP-54F28 when combined with nab-paclitaxel and gemcitabine. OMP-54F28 will be administered IV on Days 1 and 15 of each 28-day cycle. Nab-paclitaxel (125 mg/m2) and gemcitabine (1000 mg/m2) will be administered IV on Days 1, 8, and 15 of each cycle. The planned dose levels of OMP-54F28 are 3.5 mg/kg and 7.0 mg/kg.

DETAILED DESCRIPTION:
Depending on safety in this study, additional lower or intermediate dose levels may be evaluated. Depending on emerging safety data from the Phase 1a study 54F28-001 with continuing dose escalation, additional higher dose levels of OMP-54F28 may be evaluated in this study. No dose escalation of OMP-54F28 will be allowed within a dose cohort.

Once the maximum tolerated dose (MTD) or maximum administered dose (MAD) has been determined, up to 10 patients may be enrolled in the cohort-expansion phase to better characterize the safety, tolerability and PK of OMP-54F28 combined with nab-paclitaxel and gemcitabine. Up to approximately 34 patients may be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥18 years
* Histologically documented Stage IV ductal adenocarcinoma of the pancreas
* Availability of FFPE tumor tissue, either archival or obtained at study entry through fresh biopsy
* Tumor tissue from fine needle aspiration is not acceptable.
* ECOG performance status of 0 or 1
* Adequate hematologic and end-organ function
* Evaluable or measurable disease per RECIST v1.1
* For women of childbearing potential and men with partners of childbearing potential, agreement to use two effective forms of contraception

Exclusion Criteria:

* Prior therapy before Day 1 of Cycle 1 for the treatment of Stage IV pancreatic cancer
* Prior adjuvant therapy for the treatment of ductal adenocarcinoma of the pancreas
* Known hypersensitivity to any component of study treatments
* Known brain metastases, uncontrolled seizure disorder, or active neurologic disease
* Leptomeningeal disease as a manifestation of cancer
* Active infection requiring antibiotics
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known history of clinically significant liver disease, including active viral hepatitis and cirrhosis
* Significant intercurrent illness including, but not limited to, unstable angina pectoris, and cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnancy, lactation, or breastfeeding
* Known HIV infection
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Concurrent use of therapeutic warfarin
* History of interstitial lung disease, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or pulmonary hypersensitivity pneumonitis
* New York Heart Association Classification III or IV
* Known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the first dose of study treatment or anticipation of need for major surgical procedure during the course of the study
* Osteoporosis based on a T-score of <-2.5 at the left or right total hip, left or right femoral neck or lumbar spine (L1-L4) as determined by DEXA scan
* Bone metastases and one of the following:

  * Prior history of a pathologic fracture
  * Lytic lesion requiring an impending orthopedic intervention
  * Lack of treatment with a bisphosphonate or denosumab
* Treatment with a thiazolidinedione PPAR gamma inhibitor; e.g. Actos® (pioglitazone) and Avandia® (rosiglitazone)
* Active treatment with an oral or IV glucocortocoid for ≥4 weeks at a daily dose equivalent to or greater than 7.5 mg of oral prednisone
* Fasting β-CTX of >1000 pg/mL
* Metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of OMP-54F28 in combination with nab-paclitaxel and gemcitabine in patients with previously untreated Stage IV pancreatic cancer | Subjects will be treated and observed for DLT through the end of the first cycle (from Day 0 - 28)
  The maximum tolerated dose (MTD) will be determined in patients treated with gemcitabine in combination with weekly nab-paclitaxel (from Day 0 - 28)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of OMP-54F28 when administered in combination with nabpaclitaxel and gemcitabine to patients with previously untreated Stage IV pancreatic cancer | Plasma sample for Pharmacokinetics (PK) analysis to be obtained prior to the gemcitabine infusion and before nabpaclitaxel infusion from Day 0 to treatment termination
  Apparent half life, AUC, clearance, volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Colin Weekes, MD, PhD, Principal Investigator
Locations (5):
- United States (5):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee